CLINICAL TRIAL: NCT01827033
Title: Effects of Meditation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The Principal Investigator is leaving Johns Hopkins.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Miriam Mintzer, Associate Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00082735
Record Dates: First submitted 2013-03-29; First posted 2013-04-09 (Estimated); Last update posted 2015-09-16 (Estimated); Status verified 2013-11

CONDITIONS: Meditation Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- meditation training (Other)
  Interventions: Behavioral: meditation training

INTERVENTIONS:
Behavioral: meditation training

SUMMARY:
This research is being done to learn about the effects of doing meditation (sitting quietly and concentrating) on people's ability to pay attention and be relaxed.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-55
* currently enrolled in methadone maintenance program

Exclusion Criteria:

* history of: a severe medical or psychiatric condition (except substance abuse; e.g., schizophrenia); brain trauma affecting cognitive functioning
* prior experience with meditation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2013-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
computerized attention task | within 1 week after training
  discrimination score on the continuous performance task

SECONDARY OUTCOMES:
stress questionnaires | within 1 week after training
mindfulness questionnaire | within 1 week after training

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Z Mintzer, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- BPRU, Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States